CLINICAL TRIAL: NCT02442908
Title: A 12-Week, Randomised, Placebo Controlled, Multi-Centre, Parallel Group Study Assessing the Safety and Tolerability of Nutrifriend Cachexia (Non-Complete Dietary Formula) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Pilot Study of Safety and Tolerability of Nutrifriend Cachexia in COPD Cachexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smartfish AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SF-K002
Record Dates: First submitted 2015-05-07; First posted 2015-05-13 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: COPD; Cachexia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NF Cachexia (Experimental): Nutrifriend Cachexia, an Omega-3 enriched fruit juice (non complete dietary formula).
  Interventions: Dietary Supplement: Nutrifriend Cachexia
- Placebo (Placebo Comparator): An isocaloric placebo comparator
  Interventions: Dietary Supplement: Isocaloric placebo

INTERVENTIONS:
Dietary Supplement: Nutrifriend Cachexia — 2 daily for 12 weeks
  Other Names: NFCax
  Arms: NF Cachexia
Dietary Supplement: Isocaloric placebo — 2 daily for 12 weeks
  Other Names: Placobo
  Arms: Placebo

SUMMARY:
SF-K002 is a pilot study in patients with moderate to severe COPD suffering from involuntary weight loss. The study is 12 weeks, double-blinded, placebo controlled and the main objective is to study the safety and tolerability of Nutrifriend Cachexia.

DETAILED DESCRIPTION:
This study is a 12-week, randomised, parallel group, placebo controlled, multi-centre study. The primary objective is to evaluate the safety and tolerability of Nutrifriend Cachexia in patients with COPD. The secondary objectives of the study are to evaluate effects on body composition, muscle function, daily activity, inflammation, lung function, compliance, appetite and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years
* Moderate to severe COPD patients with forced expiratory volume (FEV1) of 30-60%
* Involuntary weight loss <10%
* 18 kg/m2 ≤ BMI ≤ 32 kg/m2

Exclusion Criteria:

* Exacerbation of COPD within 3 months prior to screening
* Treatment with oral corticosteroids (>5 mg/day) within 3 months prior to screening
* Treatment with anabolic steroids within 3 months prior to screening
* Current oxygen treatment or home ventilation therapy
* Change in smoking habits during the previous 6 months
* Major changes in COPD maintenance treatment within 3 months prior to screening
* Other cachectic disorders such as cancer, renal or hepatic disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by (adverse events, concomitant medication and laboratory markers) of Nutrifriend Cachexia in patients with COPD | 12 weeks

SECONDARY OUTCOMES:
Body composition assessed by fat mass and lean body mass (LBM) | 12 weeks
Body composition assessed by weight, BMI and waist & calf circumference | 12 weeks
Function assessed by 6 minute walking test | 12 weeks
Function assessed by grip strength | 12 weeks
Function assessed by walking distance | 12 weeks
Inflammation | 12 weeks
  IL-6, IL-8, TNF-alpha, CRP
Metabolic markers | 12 weeks
  Glucose, insulin, cholesterol
QoL assessed by COPD Assessment Test (CAT) | 12 weeks
QoL assessed by COPD Clinical Questionnaire (CCQ) | 12 weeks
QoL assessed by St. George Respiratory Questionnaire for COPD patients (SGRQ C) | 12 weeks
QoL assessed by Functional Assessment of Anorexia/Cachexia Therapy (FAACT) questionnaire | 12 weeks
QoL assessed by Nutrition Appetite Questionnaire (CNAQ) | 12 weeks
Compliance assessed by Drinks consumed | 12 weeks
Compliance assessed by vitamin D levels | 12 weeks
Compliance assessed by Omega-3 incorporation | 12 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - Ladulaas kliniska studier, Borås
  - Pharmasite, Helsingborg
  - Pharmasite, Malmo
  - A+ Science City Site, Stockholm

REFERENCES:
- [Background] Calder PC, Laviano A, Lonnqvist F, Muscaritoli M, Ohlander M, Schols A. Targeted medical nutrition for cachexia in chronic obstructive pulmonary disease: a randomized, controlled trial. J Cachexia Sarcopenia Muscle. 2018 Feb;9(1):28-40. doi: 10.1002/jcsm.12228. Epub 2017 Sep 10. PMID 28891198